CLINICAL TRIAL: NCT07129330
Title: Role and Mechanisms of RSPO3/SDC-1 Pathway Dysregulation in Impaired Alveolar Epithelial Repair Post-ARDS in Older Adults
Brief Title: RSPO3/SDC-1 Pathway Dysfunction in Alveolar Repair After ARDS in Older Adults
Status: Not yet recruiting | Type: Observational
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Lai Jiang, 021-25077820, Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Other Study IDs: XHEC-C-2025-167-1
Record Dates: First submitted 2025-08-12; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Acute Respiratory Distress Syndrome (ARDS); Age-related Impaired Alveolar Epithelial Repair
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- ARDS
  Interventions: Procedure: Blood and Saliva
- NON_ARDS
  Interventions: Procedure: Blood and Saliva
- AGED
  Interventions: Procedure: RSPO3/SDC-1 pathway profiling assay
- YOUNG
  Interventions: Procedure: RSPO3/SDC-1 pathway profiling assay

INTERVENTIONS:
Procedure: RSPO3/SDC-1 pathway profiling assay — Peripheral Blood: 5 mL collected into EDTA tubes; PBMCs isolated within 2 h for RT-qPCR analysis of RSPO3/SDC-1 mRNA and sandwich ELISA quantification of protein levels.
  Saliva: 2-3 mL unstimulated saliva naturally expectorated into sterile tubes, kept at 4 °C and processed within 2 h (centrifuged, aliquoted) before -80 °C storage Subcutaneous Fat: 100-200 mg obtained during elective procedures, preserved in RNAlater at 4 °C for 24 h, then frozen at -80 °C 3D Alveolar Organoid Assay: Lung tissue-derived organoids are cultured in Matrigel and treated ex vivo with recombinant RSPO3 or SDC-1 neutralizing antibody; epithelial repair is assessed over 7 days by Ki-67 immunostaining and wound-closure measurement
  Groups: AGED; YOUNG
Procedure: Blood and Saliva — Peripheral Blood: 5 mL collected into EDTA tubes; PBMCs isolated within 2 h for RT-qPCR analysis of RSPO3/SDC-1 mRNA and sandwich ELISA quantification of protein levels.
  Saliva: 2-3 mL unstimulated saliva naturally expectorated into sterile tubes, kept at 4 °C and processed within 2 h (centrifuged, aliquoted) before -80 °C storage
  Groups: ARDS; NON_ARDS

SUMMARY:
Acute respiratory distress syndrome (ARDS) is a serious lung condition in which fluid builds up in the air sacs, making it hard to breathe and often requiring intensive care. Older adults fare worse because their lung-lining cells lose the ability to heal properly after injury This study will explore two key molecules-RSPO3 and Syndecan-1 (SDC-1)-that normally help alveolar (air-sac) cells regenerate. We will collect small blood samples from ARDS patients and, when patients undergo elective lung surgery, tiny pieces of healthy lung tissue. In the lab, we will also grow three-dimensional "lung organoids" from these samples to see how boosting or blocking RSPO3/SDC-1 affects cell repair

Our goals are to:

Measure RSPO3/SDC-1 activity alongside inflammatory markers (e.g., IL-6, TNF-α) to understand their roles in age-related repair failure.

Build an integrated platform for early diagnosis, disease monitoring, and treatment evaluation in older ARDS patients.

Identify molecular targets that could lead to new therapies, helping older adults recover lung function more effectively.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of acute respiratory distress syndrome (ARDS) according to the Berlin Definition Age ≥ 65 years at enrollment First diagnosis of ARDS made within 24 hours prior to study entry Receiving either spontaneous (non-invasive) breathing support or invasive mechanical ventilation

Exclusion Criteria:

Coexisting severe cardiac, hepatic or renal failure (NYHA Class III-IV) Active pulmonary infection (e.g. pneumonia or lung abscess) Significant coagulation disorders Receipt of any cytokine-based therapy within the past 3 months Participation in another interventional clinical study within the past 3 months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: ARDS Group: 500 adult patients with acute respiratory distress syndrome, enrolled across five age brackets (20-30, 30-40, 50-60, 70-80, and > 80 years), with 100 participants per stratum Lung Resection Control Group: 500 patients undergoing elective lobectomy for non-infectious pulmonary conditions (e.g., lung tumors, interstitial lung disease), matched by age bracket and size to the ARDS cohort
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2029-12-30 (Estimated)

PRIMARY OUTCOMES:
Correlation Between Peripheral Blood RSPO3/SDC-1 Pathway Activity and Alveolar Epithelial Injury Marker Levels | Baseline (within 24 hours of ARDS diagnosis)
  Quantify RSPO3 and Syndecan-1 expression in peripheral blood (by RT-qPCR and ELISA) and measure alveolar injury biomarkers (SP-A, SP-D) in serum. Calculate Pearson or Spearman correlation coefficients between RSPO3/SDC-1 levels and SP-A/SP-D concentrations in elderly ARDS patients at baseline.

SECONDARY OUTCOMES:
Effect of RSPO3/SDC-1 Pathway Modulation on Alveolar Organoid Repair Capacity | Within 14 days of organoid establishment
  Assess lung organoid epithelial repair by measuring (1) percentage of Ki-67-positive cells and (2) wound-closure area in 3D alveolar organoid cultures treated with recombinant RSPO3 protein or SDC-1 neutralizing antibody versus untreated controls.

OTHER OUTCOMES:
Diagnostic Performance of the RSPO3/SDC-1-Based Integrated Platform | Upon completion of all sample processing (estimated by study end)
  Evaluate the multi-marker platform combining RSPO3/SDC-1 activity and inflammatory cytokines (IL-6, TNF-α) by calculating AUC, sensitivity, specificity, PPV, and NPV for predicting impaired alveolar repair in elderly ARDS patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Xinhua hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No